CLINICAL TRIAL: NCT00040027
Title: Thymosin Plus PEG-Interferon in Non-Cirrhotic Hepatitis C Patients Who Did Not Respond to Interferon or Interferon Plus Ribavirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ta1-CHC-2K0803a
Record Dates: First submitted 2002-06-18; First posted 2002-07-04 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
Keywords: hepatitis C; hepatitis C, chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Thymalfasin; peginterferon alfa-2a

INTERVENTIONS:
Drug: thymalfasin (thymosin alpha 1) + PEGinterferon alfa-2a
Drug: placebo + PEGinterferon alfa-2a

SUMMARY:
Chronic hepatitis C infection is one of the leading causes of chronic liver disease in the United States. Approximately one-third of patients with hepatitis C infection develop cirrhosis of the liver, which can lead to liver failure or liver cancer. The current treatment for hepatitis C infection in previously untreated patients is successful in only about half of patients. There is no established therapy for non-responders.

This is a randomized, double-blinded, multicenter trial to determine the effectiveness of thymosin alpha 1 (thymalfasin) 1.6 mg twice weekly plus PEGinterferon alfa-2a 180 ug/wk compared to placebo plus PEGinterferon alfa-2a in adults with chronic hepatitis C without cirrhosis who are non-responders to previous treatment with interferon or interferon plus ribavirin. The definition of non-response requires a positive HCV RNA test at the end of a course of at least 12 weeks of therapy. Patients will receive treatment for 12 months, and will be followed-up for a further 6 months after the end of therapy.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent.
* Age over 18 years old.
* Presence of HCV RNA measured by qualitative PCR.
* Nonresponder to a previous course of therapy with either IFN alone or IFN plus ribavirin. The patient must have been treated for at least 12 weeks.
* Washout period of at least 6 months from previous therapy with IFN alone or IFN plus Ribavirin.
* Liver biopsy consistent with chronic hepatitis C within the last 12 months before treatment starts, and at least 6 months after the end of the prior failed therapy.
* No clinical or histological evidence of cirrhosis (METAVIR fibrosis score 0 to 3).
* Compensated liver disease with prothrombin time prolonged less than 3 seconds over control, serum albumin stable and within normal limits, total bilirubin < 2 mg/dl, and no history of hepatic encephalopathy, esophageal varices or ascites.
* Ultrasound, CT scan, or MRI of the liver within 3 months of entry negative for HCC.
* Hematocrit > 30%, platelet count > 100 x 109/L, WBC > 3 x 109/L, and polymorphonuclear white cell count > 1.5 x 109/L.
* Adequate renal function as demonstrated by serum creatinine level < 2.0 mg/dL.
* Normal TSH or adequately controlled thyroid function.
* If the patient is a woman, she is using a definitive method of birth control in consultation with her physician, or is surgically sterile or post-menopausal.

Exclusion criteria:

* Use of systemic corticosteroids within 6 months of entry.
* Current use of any drug known to be hepatotoxic, any drug (other than the study drugs) known to have or suspected of having therapeutic activity in hepatitis C or of any immunosuppressive drug (including corticosteroids).
* Any other liver disease including hepatitis B, hepatitis delta, alcoholic liver disease, drug-induced liver injury, primary biliary cirrhosis, sclerosing cholangitis, autoimmune hepatitis, hemochromatosis, alpha 1-antitrypsin deficiency, or Wilson's disease.
* Alpha-fetoprotein > 200 ng/mL.
* Current or past diagnosis of cirrhosis.
* Evidence of portal hypertension either by Doppler ultrasonography or gastrointestinal endoscopy.
* Decompensated liver disease based on a history of hepatic encephalopathy, esophageal varices, or ascites.
* HIV infection diagnosed by HIV seropositivity and confirmed by Western blot.
* Concomitant or prior history of malignancy other than curatively treated skin cancer or surgically cured in situ carcinoma of the cervix.
* Active infectious process other than HCV that is not of a self-limited nature (eg. TB or AIDS).
* Rheumatoid arthritis or other autoimmune disease (serum ANA > 1:160).
* Pregnancy as documented by a urine pregnancy test.
* Alcohol or intravenous drug abuse within the previous 1 year.
* Chronic use of methadone.
* Patients who are poor medical risk or who have any non-malignant systemic disease that, in the opinion of the investigator, would make it unlikely that the patient could complete the protocol.
* Patients with a history of severe depression that required either hospitalization or electroshock therapy; or depression associated with suicide attempt.
* Patients with significant pre-existing cardiac or pulmonary disease.
* Any indication that the patient would not comply with the conditions of the study protocol.
* Previous treatment with thymosin alpha 1.
* Patients with known hypersensitivity to IFNa.
* Simultaneous participation in another investigational drug study, or participation in any clinical trial involving investigational drugs with 3 months before study entry.
* Family history of intracerebral hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-04

CONTACTS AND LOCATIONS:
Locations (48):
- United States (46):
  - University of Alabama - Knollwood Physician's Group Bldg., Mobile, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Gastroenterology Associates of East Bay Medical Group, Berkeley, California
  - Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Veterans Administration Medical Center GI Section (111B), San Francisco, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Center for Digestive and Liver Health, Savannah, Georgia
  - Idaho Gastroenterology Associates, Meridian, Idaho
  - University of Chicago Hospital & Clinic, Chicago, Illinois
  - Hepatitis C Treatment Centers, Inc., Louisville, Kentucky
  - Liver Research Center - University of Louisville, Louisville, Kentucky
  - Louisiana State University Healthcare Network, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - New England Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mississippi Gastrointestinal Associates, Jackson, Mississippi
  - VAMC, Kansas City, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Bronx VA Medical Center, New York, New York
  - NY VAMC, New York, New York
  - NYU Hospitals Center, New York, New York
  - Carolinas Center for Liver Diseases, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati - College of Medicine, Cincinnati, Ohio
  - Metro Health Medical Center, GI Division, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - GI Center MidSouth, Memphis, Tennessee
  - University of Tennessee Gastroenterology, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor, VAMC, Houston, Texas
  - Metropolitan Research, Fairfax, Virginia
  - McGuire Research Institute, Richmond, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - Fundacion de Investigacion de Diego, Santurce